CLINICAL TRIAL: NCT04383145
Title: INNER-B - A Post-market Clinical Follow-up Study in Patients With Thoracoabdominal Aortic Aneurysms Treated With E-nside TAAA Multibranch Stent Graft System
Brief Title: A Study in Patients With Thoracoabdominal Aortic Aneurysm Treated With the E-nside TAAA Multibranch Stent Graft System
Acronym: INNER-B
Status: Recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: INNER-B
Record Dates: First submitted 2020-05-03; First posted 2020-05-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Vascular Aneurysm
Keywords: Thoracoabdominal; aorta; aneurysm; endovascular; repair
MeSH Terms: conditions — Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endovascular repair — Endovascular repair of thoracoabdominal aneurysm using stent grafts.

SUMMARY:
The INNER-B post-market clinical follow-up study is undertaken to evaluate the prevention of death related to a thoracoabdominal aneurysm when treated by the E-nside TAAA Multibranch Stent Graft System.

The secondary objective is to evaluate the safety and clinical performance of the device.

DETAILED DESCRIPTION:
In this study patients will be observed, who receive an E-nside TAAA Multibranch Stent Graft System for the endovascular treatment of a degenerative, atherosclerotic thoracoabdominal aortic aneurysm. The E-nside TAAA Multibranch Stent Graft will be implanted at the discretion of the treating physician.

Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with the E-nside TAAA Multibranch Stent Graft System. Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before data are being collected.

The period of data collection will be approximately 60 months from the index procedure for each patient. Source document verification will be performed on 100% of patients; data from all visits will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans will be sent to the CoreLab for independent evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 85 years old
* Patient has a degenerative, atherosclerotic thoracoabdominal aortic aneurysm
* Patient has adequate iliac/femoral access compatible with an 8.5 mm OD delivery system
* Patient's aorta has no distinct angulation in the thoracovisceral segment of the aorta ranging from 40 mm proximal to the celiac trunk to 20 mm distal to the lowest renal artery
* All target branch vessels are suitable for antegrade cannulation
* Diameter of the landing zone in each branch vessel to be treated is ≥ 5 mm
* Length of landing zone in each branch vessel to be treated is ≥ 15 mm (preferably ≥ 20 mm)
* Patient must be available for the appropriate follow-up times for the duration of the study
* Patient has signed the informed consent before implantation of the E-nside Stent Graft

Exclusion Criteria:

* Patient has allergies to materials necessary for endovascular repair (e.g. contrast media, anticoagulants or heparin, nitinol, polyester, gold, platinum-iridium)
* Patient has systemic infection or suspected systemic infection
* Patient has an infectious aneurysm
* Patient has an inflammatory aneurysm
* Patient has a ruptured aneurysm
* Patient has a traumatic aneurysm
* Patient has a symptomatic aneurysm
* Patient has an aortic dissection
* Patient has a congenital degenerative collagen disease or connective tissue disorder
* Diameter of ostium of branch vessel to be treated < 4 mm
* Patient has thrombocytopenia (platelet count < 150000/µl)
* Patient has an eGFR < 30 ml/min/1.73m2 before the enrolment
* Patient has untreated hyperthyroidism
* Patient has a malignancy (progressive, stable or partial remission) with less than one-year projected survival
* Patient had a myocardial infarction or cerebrovascular accident < 3 months ago
* Patient is planned to be treated with a chimney in the left subclavian artery
* Patient has had a previous surgical repair of descending thoracic aorta
* Patient will be treated or had been treated with a Nellix (Endologix) or Ovation (Endologix) or Altura (Lombard Medical) or Anaconda (Vascutek) stent graft
* Patient is enrolled or plans to be enrolled in another clinical study
* Patient is pregnant or breastfeeding or planning to become pregnant during the course of the study.
* Patient has a life expectancy of less than 3 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with degenerative, atherosclerotic thoracoabdominal aortic aneurysm who are scheduled for implantation of an E-nside TAAA Multibranch Stent Graft at their physician's discretion and who are eligible in accordance with the inclusion / exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of all-cause mortality in peri-operative periods (all related interventions)
Mortality | 3-6, 12, 24, 36, 60 months
  Rate of all-cause mortality
Rupture | 30-day, 3-6, 12, 24, 36, 60 months
  Rate of patients with aneurysm rupture
Major Adverse Events (MAE) | prior to discharge, 30 days, 3-6, 12, 24, 36, 60 months
  Rate of patients with major adverse events (aneurysm related death, aneurysm rupture, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke, visceral ischemia (bowel ischemia with surgery or submission to ICU or bowel necrosis with surgery or submission to ICU), new hepatic infarction, new chronic renal insufficiency/renal failure requiring dialysis, new permanent paraplegia, new permanent paraparesis, lower limb ischemia (increase in Rutherford classification) (product-related, procedure-related, aneurysm-related)
Number of intervention(s) | perioperative
  Rate of interventions in peri-operative periods (all related interventions until index procedure)
Delivery time | perioperative
  Rate of time intervals the E-nside delivery system remained in the access vessels in relation to the number of branches treated with pre-cannulation
Reintervention | 30 days, 3-6, 12, 24, 36, 60 months
  Rate of reintervention(s)
Endoleak Type Ia | 12, 24, 36, 60 months
  Rate of patients with type Ia endoleak
Endoleak Type Ib | 12, 24, 36, 60 months
  Rate of patients with type Ib endoleak
Endoleak Type Ic | 12, 24, 36, 60 months
  Rate of patients with type Ic endoleak
Endoleak Type II | 12, 24, 36, 60 months
  Rate of patients with type II endoleak
Endoleak Type III | 12, 24, 36, 60 months
  Rate of patients with type III endoleak
Endoleak Type IV | 12, 24, 36, 60 months
  Rate of patients with type IV endoleak
Endoleak of unknown origin | 12, 24, 36, 60 months
  Rate of patients with endoleak of unknown origin
Proximal intercomponent separation | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of patients with intercomponent separation at the proximal end of the E-nside stent graft > 10 mm
Distal intercomponent separation | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of patients with intercomponent separation at the distal end of the E-nside stent graft > 10 mm
Integrity | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of patients with loss of device integrity (stent fracture and tear in graft material and suture break)
Kinking | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of patients with E-nside stent graft or bridging stent graft kinking
Primary patency | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of primary patency of bridging stents
Primary patency of bridging stent of the celiac trunk | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of primary patency of the bridging stent of the celiac trunk
Primary patency of bridging stent of the superior mesenteric artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of primary patency of the bridging stent of the superior mesenteric artery
Primary patency of bridging stent of the right renal artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of primary patency of the bridging stent of the right renal artery
Primary patency of bridging stent of the left renal artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of primary patency of the bridging stent of the left renal artery
Secondary patency | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of secondary patency of bridging stents
Secondary patency of the bridging stent of the celiac trunk | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of secondary patency of the bridging stent of the celiac trunk
Secondary patency of the bridging stent of the superior mesenteric artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of secondary patency of the bridging stent of the superior mesenteric artery
Secondary patency of the bridging stent of the right renal artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of secondary patency of the bridging stent of the right renal artery
Secondary patency of the bridging stent of the left renal artery | prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of secondary patency of the bridging stent of the left renal artery
Infection | 30-day, 12, 24, 36, 60 months
  Rate of patients with stent graft infection
Primary technical success | 24 hours
  Rate of patients with primary technical success. Technical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated within 24 h after the index procedure.
  Successful introduction and deployment of the E-nside TAAA Multibranch Stent Graft in the absence of:
  Surgical conversion Mortality Reintervention Unplanned branch vessel occlusion (post-operative occlusion)
  Including:
  Secure proximal and distal fixation Patent treated branch vessels
Technical success | 24 hours
  Rate of patients with technical success. Technical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated after the index procedure.
Primary clinical success | 12, 24, 36, 60 months
  Rate of patients with primary clinical success.
  Primary clinical success is reported on an intent-to-treat basis and is reached if the following criteria are fulfilled at the time of follow-up starting at 12 months follow-up:
  Successful deployment of the endovascular devices at the intended location in the absence of:
  Death as result of aneurysm-related treatment Conversion to open repair Reintervention after index procedure Occlusion of treated branch vessels Type I or III endoleak Increasing aneurysm size Aneurysm rupture
Clinical success | 12, 24, 36, 60 months
  Rate of patients with clinical success. Clinical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated after the index procedure.
Stable aneurysm size | 12, 24, 36, 60 months
  Rate of patients with stable aneurysm size
Decreasing (< 5 mm) aneurysm size | 12, 24, 36, 60 months
  Rate of patients with decreasing aneurysm size
Increasing (> 5 mm) aneurysm size | 12, 24, 36, 60 months
  Rate of patients with increasing aneurysm size
Stent graft removal | 24 hours, prior to discharge/30 days, 12, 24, 36, 60 months
  Rate of patients with removal or failure to implant the E-nside TAAA Multibranch Stent Graft

CONTACTS AND LOCATIONS:
Overall Officials: Dittmar Böckler, Prof. Dr., Study Director — University Hospital Heidelberg
Locations (1):
- Universitätsklinikum Heidelberg, Heidelberg, Germany